CLINICAL TRIAL: NCT06961214
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study of the Efficacy and Safety of Depemokimab in Adult Participants With COPD With Type 2 Inflammation
Brief Title: Depemokimab as an Extended treatmeNt Duration Biologic in Adults With Chronic Obstructive Pulmonary Disease (COPD) and Type 2 Inflammation (ENDURA-2)
Acronym: ENDURA-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 222725; 2024-520417-41 (EudraCT Number)
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Depemokimab; GSK3511294; Eosinophilic phenotype; Chronic obstructive pulmonary disease; COPD; Moderate COPD; Severe COPD; Uncontrolled Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD); Exacerbations; Placebo; Type 2 inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study neither the participants the caregivers the researchers nor the people assessing the outcomes know which treatment is being given to whom.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Depemokimab (Experimental): Participants will be administered subcutaneous (SC) injection of Depemokimab along with standard of care (SoC).
  Interventions: Drug: Depemokimab
- Placebo (Placebo Comparator): Participants will be administered placebo along with SoC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Depemokimab — Depemokimab as a sterile liquid formulation will be administered.
  Other Names: GSK3511294
  Arms: Depemokimab
Drug: Placebo — Placebo as a sterile 0.9 percent (%) sodium chloride solution will be administered
  Arms: Placebo

SUMMARY:
Depemokimab is being developed as a treatment for individuals with moderate to severe COPD. The aim of this study is to assess the efficacy and safety of depemokimab compared as an add-on medicine in participants with uncontrolled moderate to severe COPD with type 2 inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to (>=) 40 to less than or equal to (<=) 80 years of age, at the time of signing the Informed consent
* Elevated Blood Eosinophil Count (BEC)
* Moderate to severe COPD with frequent exacerbations, defined as:

  * A clinically documented history of COPD as defined by the American Thoracic Society/European Respiratory Society for at least 1 year
  * A post-bronchodilator forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) ratio of < 0.70 and a post-bronchodilator FEV1 >30 percent (%) and <= 80% predicted normal values
  * A well-documented history of at least 2 moderate or 1 severe exacerbation in the 12 months prior to screening
* COPD assessment test (CAT) score >=10 at Visit 1
* Smoking status: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years.
* Participants should be on optimized inhaler therapy, defined as inhaled corticosteroid (ICS) plus Long-acting muscarinic receptor antagonist (LAMA) plus Long-acting beta2-adrenergic receptor agonist (LABA) either as multiple inhalers or a single combination inhaler for at least 6 months prior to Screening Visit 1
* Body mass index (BMI) >=16 kilogram per square meter (kg/m^2)
* Male and eligible female participants

Exclusion Criteria:

The following subjects are excluded:

* Participants with a current or prior physician diagnosis of asthma
* Other clinically significant lung disease: The Investigator must judge that COPD is the primary diagnosis accounting for the clinical manifestations of the lung disease
* Participants with pneumonia, COPD exacerbation, or lower respiratory tract infection within the 4 weeks prior to Screening Visit 1
* Lung resection: Participants with a history of or plan for lung volume reduction surgery / endobronchial valve procedure.
* Pulmonary rehabilitation: Participants in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening Visit 1
* Continuous oxygen: Participants requiring oxygen supplementation for more than 12 hours per day
* Cor pulmonale - resulting in right heart failure, severe pulmonary hypertension
* Chronic hypercapnia requiring Non-invasive positive pressure ventilation (NIPPV) use (including Bi-Level Positive Airway Pressure [BiPAP] or Continuous Positive Airway Pressure [CPAP])
* Unstable cardiovascular disease or arrhythmia
* Parasitic Infection: Participants with a known, pre-existing parasitic infection within 6 months of Screening (Visit 1)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2029-08-21 (Estimated); Study Completion 2029-08-21 (Estimated)

PRIMARY OUTCOMES:
Annualized Rate of Moderate/Severe Exacerbations | From Baseline up to Week 104
  Moderate exacerbations are defined as clinically significant exacerbations that require treatment with oral/systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as clinically significant exacerbations that require in-patient hospitalization (i.e., greater than or equal to [>=] 24 hours) or result in death. The frequency of moderate/ severe exacerbations expressed as an annualized exacerbation rate will be evaluated.

SECONDARY OUTCOMES:
Time to First Moderate/Severe Exacerbation | From Baseline up to Week 104
  Moderate exacerbations are defined as clinically significant exacerbations that require treatment with oral/systemic corticosteroids and/or antibiotics. Severe exacerbations are defined as clinically significant exacerbations that require in-patient hospitalization (i.e., greater than or equal to [>=] 24 hours) or result in death.
Change from Baseline in St. George's Respiratory Questionnaire (SGRQ) Total Score at Week 52 | From Baseline up to Week 52
  The SGRQ total score will be measured using the SGRQ for COPD [SGRQ-C]. The SGRQ-C is a 40-item participant questionnaire designed to measure health impairment by addressing the frequency of respiratory symptoms (questions 1-7) and the participant's current state (questions 8-14). The questions are designed to be self-completed by the participant. The total score will be calculated on 0-100 rating scale and scores expressed as a percentage of overall impairment. Higher scores indicate greater impairment of health.
Change from Baseline in Evaluating Respiratory Symptoms in Chronic Obstructive Pulmonary Disease (E-RS: COPD) Total Score at Week 52 | From Baseline up to Week 52
  E-RS: COPD consists of 11 items from the 14-item Exacerbations of Chronic Pulmonary Disease Tool - Patient Reported Outcomes (EXACT) instrument. E-RS: COPD is intended to capture information related to the respiratory symptoms of COPD, i.e., breathlessness, cough, sputum production, chest congestion, and chest tightness. The E-RS: COPD has a scoring range of 0 to 40, higher scores indicate more severe symptoms.
Annualized Rate of Exacerbations Requiring Emergency Department (ED) Visit or Hospitalization | From Baseline up to Week 104
  Annualized rate of exacerbations requiring ED Visit or Hospitalization (For pooled analysis across studies 222714 and 222725) will be assessed.
Annualized Rate of Severe Exacerbations | From Baseline up to Week 104
  Severe exacerbations are defined as clinically significant exacerbations that require in-patient hospitalization (i.e., greater than or equal to [>=] 24 hours) or result in death. Annualized rate of severe exacerbations (For pooled analysis across studies 222714 and 222725) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/